CLINICAL TRIAL: NCT02645331
Title: "Remind to Move" Treatment Versus Constraint-induced Movement Therapy for Children With Hemiplegic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: "Remind to Move" Treatment Versus Constraint-induced Movement Therapy for Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20130214003
Record Dates: First submitted 2015-12-23; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Hemiplegic Cerebral Palsy; Upper Extremity Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Remind-to-move (Experimental): RTM involved a wristwatch device worn on more-affected arm which emitted sensory cueing continuously to remind the children to use the more-affected hand to engage in daily activities or complete bimanual tasks intensively, 5 hour per day, 5 days every week, for 3 consecutive weeks.
  Interventions: Behavioral: Remind-to-move
- Modified constraint induced movement therapy (mCIMT) (Active Comparator): children were encouraged to wear a customer-made volar resting splint that extended from below the elbow to the fingertips on their noninvolved hands for 5 hour daily except for toileting, writing and specific physical sports, for 3 weeks. Each child was supervised by one therapist to complete structured unimanual practice with the affected hand during the supervised session, 5 days every week, for 3 consecutive weeks.
  Interventions: Behavioral: Modified constraint induced movement therapy
- Conventional rehabilitation (Placebo Comparator): Conventional splinting, muscle strengthening, stretching, and neurodevelopmental facilitation techniques for 1hr daily, 2 day per week for 3 weeks.
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Behavioral: Remind-to-move
  Arms: Remind-to-move
Behavioral: Modified constraint induced movement therapy
  Arms: Modified constraint induced movement therapy (mCIMT)
Behavioral: Conventional rehabilitation
  Arms: Conventional rehabilitation

SUMMARY:
The aim of this study was to determine the effects of an innovative child-friendly remind-to-move treatment (RTM) treatment by comparing it with constraint-induced movement therapy (CIMT) on upper extremity outcomes in children with hemiplegic Cerebral Palsy. In an evaluator-blinded randomized controlled trial, 73 children, among of whom 20 in Manual Ability Classification System level I, 38 level II, and 15 level III, were recruited from 3 special schools and randomized to receive 75-hour RTM (n=25) and CIMT (n=24) programme over 15-weekdays, and conventional treatment (n=24). The primary outcomes were Jebsen-Taylor Hand Function Test (JTHFT) and Bruininks-Oseretsky Test of Motor Proficiency (BOTMP-II) Subtest 3 for assessing the motor efficiency at baseline, posttest, and 1- and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hemiplegic Cerebral Palsy
* Aged 5 to 16 years
* Ability to follow instructions
* Ability to grasp and release light objects, and at least 20° wrist and 10°fingers in metacarpophalangeal joints extension from full flexion for the affected hand
* Manual Activity Classification System (MACS) 19 grades I, II or III of the affected hand

Exclusion Criteria:

* Severe cognitive, visual, or auditory disorder
* Seizure and health problems not associated with cerebral palsy
* Predominant spasticity or contracture grades more than 3 of Modified Ashworth Scale 20 on wrist and finger flexors, forearm pronators and ⁄ or thumb adductors
* Receiving new pharmaceutical (i.e. botulinum toxin injections) and/or surgical interventions within 6-month before study

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Jebsen-Taylor Hand Function Test (JTHFT) | Change from Baseline at 3 weeks (plus follow up at 1 month and 3 months after training)
Bruininks-Oseretsky Test of Motor Proficiency (2nd ed.) (BOTMP-II) | Change from Baseline at 3 weeks (plus follow up at 1 month and 3 months after training)

SECONDARY OUTCOMES:
Caregiver Functional Use Survey (CFUS) | Change from Baseline at 3 weeks (plus follow up at 1 month and 3 months after training)
Ratio of movement duration on the affected hand from accelerometer | Change from Baseline at 3 weeks (plus follow up at 1 month and 3 months after training)
Active range of motion (AROM) as measured by digital goniometer | Change from Baseline at 3 weeks (plus follow up at 1 month and 3 months after training)
Power grip strength as measured by dynamometer | Change from Baseline at 3 weeks (plus follow up at 1 month and 3 months after training)

REFERENCES:
- [Background] Fong KN, Jim ES, Dong VA, Cheung HK. 'Remind to move': a pilot study on the effects of sensory cueing treatment on hemiplegic upper limb functions in children with unilateral cerebral palsy. Clin Rehabil. 2013 Jan;27(1):82-9. doi: 10.1177/0269215512448199. Epub 2012 Jul 16. PMID 22801471
- [Background] Dong AQ, Fong NK. Remind to move - A novel treatment on hemiplegic arm functions in children with unilateral cerebral palsy: A randomized cross-over study. Dev Neurorehabil. 2016 Oct;19(5):275-83. doi: 10.3109/17518423.2014.988304. Epub 2014 Dec 30. PMID 25548861